CLINICAL TRIAL: NCT03370861
Title: Immunotherapy Multi-omics Specimen Protocol A
Brief Title: How Microbes and Metabolism May Predict Skin Cancer Immunotherapy Outcomes
Acronym: MINING
Status: Terminated | Type: Observational
Why Stopped: Subject recruitment was limited severely by the 2020-2023 COVID-19 pandemic, which led this study to be closed.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, William H. McCoy IV, MD, PhD, Research Instructor of Medicine, Washington University School of Medicine
Other Study IDs: MINING
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Autoimmunity; Melanoma; Merkel Cell Carcinoma; Squamous Cell Carcinoma of the Skin; Basal Cell Carcinoma; Skin Cancer
MeSH Terms: conditions — Autoimmune Diseases; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Basal Cell; Skin Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Immunotherapy — Medications that increase the activity of the immune system.

SUMMARY:
The purpose of this research study is to examine the relationship between the microbiota (microscopic organisms) in the gut and the activity of the immune system during skin cancer immunotherapy.

DETAILED DESCRIPTION:
Details will be available upon publication.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Diagnosis of skin cancer.
* Planning to initiate or already on ANY type of immunotherapy.
* Able to provide urine and stool specimens.

Exclusion Criteria:

* Bowel resection.
* Major GI surgery in the past 5 years other than cholecystectomy and appendectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with skin cancer planning to initiate or already on ANY type of immunotherapy.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Immune-related Adverse Events (irAEs) | 2 years
  Electronic medical records will be queried for specific drug-related adverse events known as immune-related Adverse Events (irAEs) including but not limited to colitis, hypophysitis, hepatitis, pneumonitis, pancreatitis, arthritis, rash, and vitiligo.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: William H McCoy IV, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hosptial, St Louis, Missouri, United States